CLINICAL TRIAL: NCT06063629
Title: Roles of Prophylactic Subcutaneous Drain in Preventing Surgical Site Infection in Abdominal Surgery Wound Class III and IV
Brief Title: Roles of Prophylactic Subcutaneous Drain in Preventing Surgical Site Infection in Surgical Wound After Abdominal Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Savang Vadhana Memorial Hospital, Thailand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 030/2565
Record Dates: First submitted 2023-09-22; First posted 2023-10-02 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Intervention Model Description: Minimization randomization
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subcutaneous drain (Experimental): The drain will be inserted into subcutaneous layer of the surgical wound. Redivac drain will be used in this study.
  Interventions: Procedure: Subcutaneous drain
- No drain (Other): No drain will be inserted into the surgical wound in this arm.
  Interventions: Procedure: No drain

INTERVENTIONS:
Procedure: Subcutaneous drain — The drain will be inserted into subcutaneous layer of the surgical wound. Redivac drain will be used in this study.
  Arms: Subcutaneous drain
Procedure: No drain — No drain will be inserted into patients allocated to this group
  Arms: No drain

SUMMARY:
Surgical site infections (SSI) pose a common challenge in the field of surgery. Current evidence and literature do not provide clear consensus whether the use of subcutaneous drainage will help reduce the incidence of SSI in patients who underwent abdominal surgery, especially in wounds that are categorized as contaminated (class 3) or dirty/infected (class 4).

The objective of this clinical study is to compare the rate of surgical site infection in contaminated and dirty/infected surgical wounds among patients whose wounds are inserted with subcutaneous drainage and patients who are not inserted with subcutaneous drainage.

DETAILED DESCRIPTION:
This study is a randomized, controlled and open study, where participants who undergo abdominal surgery will be randomly allocated into two groups: (i) patients whose wounds are inserted with subcutaneous negative pressure drain and (ii) patients whose wounds are not inserted with subcutaneous negative pressure drain.

The participants in this study will know the details about the presence of their drain placement after the operation. If the patient was assigned to the drain group, the drain will be placed for five days or until there are no content observed in the drain. The primary outcome of this study is the occurrence of SSI, which will be tracked up to 30 days post-operation. The patient in both groups will also be evaluated by the surgeons at day 3, 5, 7, 14 and 30 post-operation for signs and complications of SSI. In situation where the patients are discharged prior to the date of evaluation, the patients will be scheduled for evaluation during the follow-up visits.

If SSI is detected in the drain group prior to removal, the drain will be removed and the patient will be treated with wet dressing combined with antibiotics. Complications of SSI will also be noted. Patient's data on demographic, medical history, clinical presentation, details of operation, and other laboratory findings will also be collected to investigate for risk factors for development of SSI between each group.

ELIGIBILITY:
Inclusion Criteria:

* Age equal or over 18 years old
* Admitted to Queen Savang Vadhana Memorial Hospital
* Receive abdominal surgery and were classified as class 3 or 4 wound

Exclusion Criteria:

* Patients who undergo operation for ostomy
* Patients who do not receive appropriate antibiotics
* Patients who undergo operation before full recover of prior operation
* Patients who undergo laparoscopic operation
* Pregnant women
* Patients who had history of prior radiation therapy at abdomen
* Patient with immunocompromised status
* Patient with chronic skin disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Rate of Surgical Site Infection (SSI) | Post operation day 3
  The rate of SSI will be compared between the drain and no drain group
Rate of Surgical Site Infection (SSI) | Post operation day 5
  The rate of SSI will be compared between the drain and no drain group
Rate of Surgical Site Infection (SSI) | Post operation day 7
  The rate of SSI will be compared between the drain and no drain group
Rate of Surgical Site Infection (SSI) | Post operation day 14
  The rate of SSI will be compared between the drain and no drain group
Rate of Surgical Site Infection (SSI) | Post operation day 30
  The rate of SSI will be compared between the drain and no drain group

SECONDARY OUTCOMES:
Length of hospital stay | Post operation day 3
  The length of hospital stay will be compared between drain and no drain group
Length of hospital stay | Post operation day 5
  The length of hospital stay will be compared between drain and no drain group
Length of hospital stay | Post operation day 7
  The length of hospital stay will be compared between drain and no drain group
Length of hospital stay | Post operation day 14
  The length of hospital stay will be compared between drain and no drain group
Length of hospital stay | Post operation day 30
  The length of hospital stay will be compared between drain and no drain group